CLINICAL TRIAL: NCT04873739
Title: Anterior Segment Optical Coherence Tomography Study of Cornea and Tear Film Parameters in Systemic Lupus Erythematous Patients
Brief Title: AS-OCT Study of Cornea and Tear Film Parameters in SLE Patients
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Farouk Sayed Othman Abelkader, Principal Investigator, Minia University
Other Study IDs: Anterior segment OCT in SLE
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2021-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: anterior segment optical coherence tomography; tear film; dry eye; systemic lupus erythematous
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 20 patients SLE with dry eye: Anterior segment OCT for SLE patients with dry eye
  Interventions: Diagnostic Test: Anterior Segment OCT
- 30 patients SLE without dry eye: Anterior segment OCT for SLE patients without dry eye
  Interventions: Diagnostic Test: Anterior Segment OCT
- 50 normal subjects as control group of similar age and gender: Anterior segment OCT for normal subjects
  Interventions: Diagnostic Test: Anterior Segment OCT

INTERVENTIONS:
Diagnostic Test: Anterior Segment OCT — AS-OCT for SLE patients with dry eye, SLE patients without dry eye and compare them with normal subjects.

SUMMARY:
The aim of thie study to assess tear film parameters such as tear meniscus height (TMH), tear meniscus area (TMA), and tear meniscus depth (TMD). In addition, corneal pachymetry and epithelial thickness maps in SLE patients and compared to healthy subjects of similar age and gender.

DETAILED DESCRIPTION:
Systemic lupus erythematous (SLE) is a relapsing and remitting autoimmune connective tissue disorder that can affect many organs such as skin, joints, kidneys, eye, and brain (1) . SLE has a global prevalence of 0.3 to 23.2 cases per 100,000. Women are more likely than men to develop the disease. Four out of the following 11 diagnostic criteria are sufficient for the diagnosis of SLE, malar rash, discoid rash, oral ulcers, non-erosive arthritis, serositis, photosensitivity, renal disorder, neurological disorder, hematological disorder, immunological disorder, and presence of antinuclear antibodies. (2,3)

Ocular manifestations occur in about one third of SLE patients with keratoconjunctivitis sicca being the most common manifestation which is characterized by decreased tear film aqueous layer. Scleritis, retinal vasculitis (which is often associated with CNS lupus), and papillitis are considered as the most serious ocular manifestations. (4)

Corneal involvement in SLE affects the superficial epithelium, resulting in superficial punctate keratitis, which is believed to be caused by Sjögren's syndrome (SS). However, some cases of non-infiltrative and infiltrative peripheral ulcerative keratitis have been identified (5) .

Schirmer's test and fluorescein breakup time test (FBUT) are two common clinical tests used to analyze tear film. (6,7) Using an in vivo, non- contact technique, anterior segment optical coherence tomography (AS- OCT) is now used to image the tear film, measure the lower tear film height and area, measure corneal thickness (pachymetry), and measure surface epithelial thickness. (8,9)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old..
2. Patients with SLE diagnosed by a rheumatologist with no ocular involvement upon clinical examination

Exclusion Criteria:

* 1. Patients with history of intraocular surgery as cataract surgery ,retinal detachment surgery, anti-glucoma surgery.

  2. Patients with history of any corneal refractive surgery as LASIK, PRK. 3. Patients with significant media opacity as corneal opacity, cataract. 4. Patients with ocular diseases as glaucoma, uveitis. 5. Patients with any retinal affection as pathological myopia, macular hole, age related macular degeneration and retinal vascular occlusion.

  6. Patients with systemic diseases as diabetes mellitus, hypertension, abnormal kidney function.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents of Minia Governorate diagnosed with SLE and healthy one
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Measurement of Tear meniscus | 3 months
  to measure lower tear meniscus height and area and depth with AS-OCT and comparing results between 3 groups; SLE patients with dry eye, SLE patients without dry eye and normal subjects.
Measurement of corneal structural changes | 3 months
  To measure corneal Thickness, epithelial thickness and stromal thickness using AS-OCT comparing results between 3 groups; SLE patients with dry eye, SLE patients without dry eye and normal subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelkader, Doctor, Principal Investigator — Minia University Hospital; Mohamed Salah, Doctor, Study Director — Minia University Hospital; Mohamed Hamid, Doctor, Study Director — Minia University Hospital
Locations (1):
- Minia university hospital, Minya, Egypt

REFERENCES:
- [Background] Palejwala NV, Walia HS, Yeh S. Ocular manifestations of systemic lupus erythematosus: a review of the literature. Autoimmune Dis. 2012;2012:290898. doi: 10.1155/2012/290898. Epub 2012 Jul 2. PMID 22811887
- [Background] Rees F, Doherty M, Grainge MJ, Lanyon P, Zhang W. The worldwide incidence and prevalence of systemic lupus erythematosus: a systematic review of epidemiological studies. Rheumatology (Oxford). 2017 Nov 1;56(11):1945-1961. doi: 10.1093/rheumatology/kex260. PMID 28968809
- [Background] Yu C, Gershwin ME, Chang C. Diagnostic criteria for systemic lupus erythematosus: a critical review. J Autoimmun. 2014 Feb-Mar;48-49:10-3. doi: 10.1016/j.jaut.2014.01.004. Epub 2014 Jan 21. PMID 24461385
- [Background] Read RW. Clinical mini-review: systemic lupus erythematosus and the eye. Ocul Immunol Inflamm. 2004 Jun;12(2):87-99. doi: 10.1080/09273940490895308. PMID 15512979
- [Background] Benitez del Castillo JM, Wasfy MA, Fernandez C, Garcia-Sanchez J. An in vivo confocal masked study on corneal epithelium and subbasal nerves in patients with dry eye. Invest Ophthalmol Vis Sci. 2004 Sep;45(9):3030-5. doi: 10.1167/iovs.04-0251. PMID 15326117
- [Background] Kanellopoulos AJ, Aslanides IM, Asimellis G. Correlation between epithelial thickness in normal corneas, untreated ectatic corneas, and ectatic corneas previously treated with CXL; is overall epithelial thickness a very early ectasia prognostic factor? Clin Ophthalmol. 2012;6:789-800. doi: 10.2147/OPTH.S31524. Epub 2012 May 23. PMID 22701079
- [Background] Nguyen P, Huang D, Li Y, Sadda SR, Ramos S, Pappuru RR, Yiu SC. Correlation between optical coherence tomography-derived assessments of lower tear meniscus parameters and clinical features of dry eye disease. Cornea. 2012 Jun;31(6):680-5. doi: 10.1097/ICO.0b013e3182261577. PMID 22378111
- [Background] Li Y, Tan O, Brass R, Weiss JL, Huang D. Corneal epithelial thickness mapping by Fourier-domain optical coherence tomography in normal and keratoconic eyes. Ophthalmology. 2012 Dec;119(12):2425-33. doi: 10.1016/j.ophtha.2012.06.023. Epub 2012 Aug 20. PMID 22917888